CLINICAL TRIAL: NCT07384078
Title: HIFU vs. CRYO - High Intensity Focused Ultrasound vs. Cryotherapy in the Treatment of Basal Cell Carcinomas and Bowen's Disease - a Randomized Controlled Trial
Brief Title: High Intensity Focused Ultrasound vs. Cryotherapy in the Treatment of Basal Cell Carcinomas and Bowen's Disease in Adults
Acronym: HIFUvsCRYO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jussi Salonen (Other)
Collaborators: HUS Skin and Allergy Hospital (Other)
Responsible Party: Sponsor-Investigator, Jussi Salonen, Clinical Investigator, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUS/6520/2025
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Superficial Basal Cell Carcinoma; Nodular Basal Cell Carcinoma; Bowen's Disease; BCC; BD
Keywords: HIFU; cryo; cryotherapy; high intensity focused ultrasound; basal cell carcinoma; Bowen's disease; superficial basal cell carcinoma; nodular basal cell carcinoma; non-surgical treatment
MeSH Terms: conditions — Bowen's Disease; Carcinoma, Basal Cell | interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sBCC (Experimental): Superficial basal cell carcinoma
  Interventions: Device: High Intensity Focused Ultrasound; Procedure: Cryotherapy
- nBCC (Experimental): Nodular basal cell carcinoma
  Interventions: Device: High Intensity Focused Ultrasound; Procedure: Cryotherapy
- BD (Experimental): Bowen's disease
  Interventions: Device: High Intensity Focused Ultrasound; Procedure: Cryotherapy

INTERVENTIONS:
Device: High Intensity Focused Ultrasound — High intensity focused ultrasound
  Other Names: HIFU
Procedure: Cryotherapy — Liquid nitrogen cryotherapy
  Other Names: CRYO

SUMMARY:
This prospective, randomized, controlled, and single-blinded non-inferiority clinical trial compare the efficacy and tolerability of high intensity focused ultrasound (HIFU) to standard cryotherapy in the treatment of low-risk basal cell carcinomas (BCCs) and Bowen's disease (BD) in adults. The main questions it aims to answer are:

* Is HIFU an efficient treatment option for BCCs and BD?
* What medical problems do participants get after HIFU?

Researchers will compare HIFU to standard cryotherapy with liquid nitrogen to see if the ultrasound works to treat these local and low-risk non-melanosytic skin cancers.

Participants will:

* Be treated either with HIFU (intervention) or cryotherapy (control).
* Visit the clinic 4 weeks, 1-, 3- and 5 years after the treatment for check-ups, tests and survey questions.

DETAILED DESCRIPTION:
Low-risk BCCs and BD are both local keratinocyctic skin cancers with increasing prevalence and they cause a rising burden to the health care system. In this study we assess the efficacy of HIFU compared to liquid nitrogen cryotherapy between years 2025-2030.

Alltogether 294 patients are recruited based on referrals or from patients attending the clinic, with histologically confirmed BD, superficial BCC or nodular BCC located between neck and knees. 98 tumors of each aforementioned subtypes will be recruited and randomized with 1:1 ratio to HIFU and CRYO - groups. Follow-up appointments are 4 weeks, 1-, 3- and 5 years post treatment.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older at the time of informed consent
* ability to give informed consent and comply with the treatment protocol and follow-up plan
* study lesion located between neck and knees
* one of following histologically confirmed diagnosis: Superficial BCC with maximum diameter of 2.0 cm / Nodular BCC with max. diameter of 1.5 cm / BD with max. diameter of 2.0 cm

Exclusion Criteria:

* Study lesion location in face, head, genitals, hands, or below the knee
* Clinical/dermoscopical/histological feature for high-risk/aggressive BCC
* Clinical/histological sign for hypertrophic BD
* Clinical/dermoscopical/histological feature for Squamous cell carcinoma
* Gorlin Golz syndrome
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment efficacy | From treatment to the end of follow up at 5 years
  Histologically confirmed recurrence-free survival assessed at 1, 3 and 5 years after treatment. Recurrence during follow up: Yes/no.

SECONDARY OUTCOMES:
Pain during treatment assessed by NRS | Pain during treatment procedure on treatment visit
  Zero is equivalent to no pain and 10 indicates the worst possible pain
Pain after treatment previous 4 weeks NRS | From treatment to the control visit at 4 weeks
  Zero is equivalent to no pain and 10 indicates the worst possible pain
Post treatment reactions assessed by both observer and patient | From treatment to the control visit at 4 weeks
  Yes/no: crust, ulceration, erosion, erythema, oozing, infection
Healing result assessed by both observer and patient | From treatment to the control visit at 4 weeks
  Healed (defined as no ulcer/crust left)? Yes/no
Healing time assessed by patient. How many weeks ago? | From treatment to the control visit at 4 weeks
  If defined as healed by the patient.
Cosmetic outcome assessed by both observer and the patient | From 1 year control to the end of follow up at 5 years
  Poor/fair/goof/excellent
Patient satisfaction inquiry, modified 6 questions | From 1 year control to the end of follow up at 5 years
  Patients will be asked about an overall satisfaction with the provided treatment, recommendation of the received treatment to other patients, readiness to undergo the same treatment again and post-treatment recovery and its impact on daily life. Answers will be evaluated with a modified NRS-scale from 0 to 10
Scarring after treatment POSAS 2.0 | From 1 year control to the end of follow up at 5 years
  Patient and Observer Scar Assessment Scale (POSAS 2.0)
Other adverse events related to the given treatment | From treatment visit to the end of follow up at 5 years
  Separate inquiry of adverse events

OTHER OUTCOMES:
Treatment costs | From treatment to the control at 4 weeks
  Time and resources required on treatment, cost effectiveness analysis

CONTACTS AND LOCATIONS:
Overall Officials: Sari Koskenmies, Head of Department, Principal Investigator — Helsinki University Hospital, Skin and Allergy Hospital, Dermatologic procedure unit
Locations (1):
- HUS Iho- ja allergiasairaala, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
The informed consent obtained from participants does not include permission for sharing individual-level data with external researchers. Also, data sharing is restricted due to institutional and contractual agreements that do not permit external distribution of individual-level data.

REFERENCES:
- [Background] The Finnish Cancer Registry; Syöpätilastosovellus. Vuosiraportti 2023. [Internet]. [cited 2025 Nov 19]. Available from: https://syoparekisteri.fi/tilastot/tautitilastot/
- [Background] Schlessinger DI, Reynolds KA, Dirr MA, Ibrahim SA, Yanes AF, Lazaroff JM, Godinez-Puig V, Chen BR, Kurta AO, Cotseones JK, Chiren SG, Furlan KC, Iyengar S, Behshad R, DeHoratius DM, Denes P, Drucker AM, Dzubow LM, Etzkorn JR, Harwood CA, Kim JYS, Lawrence N, Lee EH, Lissner GS, Marghoob AA, Matin RN, Mattox AR, Mittal BB, Thomas JR, Zhou XA, Zloty D, Schmitt J, Kirkham JJ, Armstrong AW, Basset-Seguin N, Billingsley EM, Bordeaux JS, Brewer J, Brown M, Brown M, Collins SAB, Fargnoli MC, De Azevedo SJ, Dummer R, Eggermont A, Goldman GD, Haedersdal M, Hale EK, Hanlon A, Harms KL, Huang CC, Hurst EA, In GK, Kelleners-Smeets N, Kheterpal M, Leshin B, Mcdonald M, Miller SJ, Miller A, Mostow EN, Trakatelli M, Nehal KS, Ratner D, Rogers H, Sarin KY, Soon SL, Stasko T, Storrs PA, Tagliaferri L, Vidimos AT, Wong SL, Yu SS, Zalaudek I, Zeitouni NC, Zitelli JA, Poon E, Sobanko JF, Cartee TV, Maher IA, Alam M. Development of a core outcome set for basal cell carcinoma. J Am Acad Dermatol. 2022 Sep;87(3):573-581. doi: 10.1016/j.jaad.2022.04.059. Epub 2022 May 10. PMID 35551965
- [Background] Hansen JP, Drake AL, Walling HW. Bowen's Disease: a four-year retrospective review of epidemiology and treatment at a university center. Dermatol Surg. 2008 Jul;34(7):878-83. doi: 10.1111/j.1524-4725.2008.34172.x. PMID 18363722
- [Background] Wang I, Bendsoe N, Klinteberg CA, Enejder AM, Andersson-Engels S, Svanberg S, Svanberg K. Photodynamic therapy vs. cryosurgery of basal cell carcinomas: results of a phase III clinical trial. Br J Dermatol. 2001 Apr;144(4):832-40. doi: 10.1046/j.1365-2133.2001.04141.x. PMID 11298545
- [Background] Basset-Seguin N, Ibbotson SH, Emtestam L, Tarstedt M, Morton C, Maroti M, Calzavara-Pinton P, Varma S, Roelandts R, Wolf P. Topical methyl aminolaevulinate photodynamic therapy versus cryotherapy for superficial basal cell carcinoma: a 5 year randomized trial. Eur J Dermatol. 2008 Sep-Oct;18(5):547-53. doi: 10.1684/ejd.2008.0472. Epub 2008 Aug 8. PMID 18693158
- [Background] Seppä K, Lappi-Heikkinen S, Johansson S, Malila N, Pitkäniemi J. SYÖPÄ 2023 Tilastoraportti Suomen syöpätilanteesta. Suomen Syöpäyhdistys, Helsinki 2025.
- [Background] Keratinocyte Cancer Clinical Guidelines | Cancer Council [Internet]. [cited 2025 Nov 19]. Available from: https://www.cancer.org.au/clinical-guidelines/skin-cancer/keratinocyte-cancer
- [Background] Telfer NR, Colver GB, Morton CA; British Association of Dermatologists. Guidelines for the management of basal cell carcinoma. Br J Dermatol. 2008 Jul;159(1):35-48. doi: 10.1111/j.1365-2133.2008.08666.x. PMID 18593385
- [Background] Newlands C, Currie R, Memon A, Whitaker S, Woolford T. Non-melanoma skin cancer: United Kingdom National Multidisciplinary Guidelines. J Laryngol Otol. 2016 May;130(S2):S125-S132. doi: 10.1017/S0022215116000554. PMID 27841126
- [Background] Work Group; Invited Reviewers; Kim JYS, Kozlow JH, Mittal B, Moyer J, Olencki T, Rodgers P. Guidelines of care for the management of basal cell carcinoma. J Am Acad Dermatol. 2018 Mar;78(3):540-559. doi: 10.1016/j.jaad.2017.10.006. Epub 2018 Jan 10. PMID 29331385
- [Background] Bichakjian CK, Olencki T, Aasi SZ, Alam M, Andersen JS, Berg D, Bowen GM, Cheney RT, Daniels GA, Glass LF, Grekin RC, Grossman K, Higgins SA, Ho AL, Lewis KD, Lydiatt DD, Nehal KS, Nghiem P, Olsen EA, Schmults CD, Sekulic A, Shaha AR, Thorstad WL, Tuli M, Urist MM, Wang TS, Wong SL, Zic JA, Hoffmann KG, Engh A. Basal Cell Skin Cancer, Version 1.2016, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2016 May;14(5):574-97. doi: 10.6004/jnccn.2016.0065. PMID 27160235
- [Background] Peris K, Fargnoli MC, Kaufmann R, Arenberger P, Bastholt L, Seguin NB, Bataille V, Brochez L, Del Marmol V, Dummer R, Forsea AM, Gaudy-Marqueste C, Harwood CA, Hauschild A, Holler C, Kandolf L, Kellerners-Smeets NWJ, Lallas A, Leiter U, Malvehy J, Marinovic B, Mijuskovic Z, Moreno-Ramirez D, Nagore E, Nathan P, Stratigos AJ, Stockfleth E, Tagliaferri L, Trakatelli M, Vieira R, Zalaudek I, Garbe C; EADO"A, EDF"B, ESTRO"C, UEMS"D and EADV"E. European consensus-based interdisciplinary guideline for diagnosis and treatment of basal cell carcinoma-update 2023. Eur J Cancer. 2023 Oct;192:113254. doi: 10.1016/j.ejca.2023.113254. Epub 2023 Jul 28. PMID 37604067
- [Background] Skin Cancer Foundation. Skin Cancer Information [Internet]. [cited 2025 Nov 19]. Available from: https://www.skincancer.org/skin-cancer-information/
- [Background] Soegaard S, Aarup V, Serup J, Bove T, Zawada T, Jessen A, Poli M. High-frequency (20 MHz) high-intensity focused ultrasound system for dermal intervention: A 12-week local tolerance study in minipigs. Skin Res Technol. 2020 Mar;26(2):241-254. doi: 10.1111/srt.12786. Epub 2019 Sep 20. PMID 31541524
- [Background] Bove T, Zawada T, Serup J, Jessen A, Poli M. High-frequency (20-MHz) high-intensity focused ultrasound (HIFU) system for dermal intervention: Preclinical evaluation in skin equivalents. Skin Res Technol. 2019 Mar;25(2):217-228. doi: 10.1111/srt.12661. Epub 2019 Jan 8. PMID 30620418
- [Background] Kim M, Jung NY, Park CK, Chang WS, Jung HH, Chang JW. Comparative Evaluation of Magnetic Resonance-Guided Focused Ultrasound Surgery for Essential Tremor. Stereotact Funct Neurosurg. 2017;95(4):279-286. doi: 10.1159/000478866. Epub 2017 Aug 16. PMID 28810261
- [Background] Lang BH, Wu ALH. High intensity focused ultrasound (HIFU) ablation of benign thyroid nodules - a systematic review. J Ther Ultrasound. 2017 May 17;5:11. doi: 10.1186/s40349-017-0091-1. eCollection 2017. PMID 28523127
- [Background] Peek MCL, Wu F. High-intensity focused ultrasound in the treatment of breast tumours. Ecancermedicalscience. 2018 Jan 10;12:794. doi: 10.3332/ecancer.2018.794. eCollection 2018. PMID 29434660
- [Background] Lamsam L, Johnson E, Connolly ID, Wintermark M, Hayden Gephart M. A review of potential applications of MR-guided focused ultrasound for targeting brain tumor therapy. Neurosurg Focus. 2018 Feb;44(2):E10. doi: 10.3171/2017.11.FOCUS17620. PMID 29385922
- [Background] Barile A, Arrigoni F, Zugaro L, Zappia M, Cazzato RL, Garnon J, Ramamurthy N, Brunese L, Gangi A, Masciocchi C. Minimally invasive treatments of painful bone lesions: state of the art. Med Oncol. 2017 Apr;34(4):53. doi: 10.1007/s12032-017-0909-2. Epub 2017 Feb 24. PMID 28236103
- [Background] Quinn SD, Gedroyc WM. Thermal ablative treatment of uterine fibroids. Int J Hyperthermia. 2015 May;31(3):272-9. doi: 10.3109/02656736.2015.1010608. Epub 2015 Mar 27. PMID 25815582
- [Background] Ellens NP, Partanen A. Preclinical MRI-Guided Focused Ultrasound: A Review of Systems and Current Practices. IEEE Trans Ultrason Ferroelectr Freq Control. 2017 Jan;64(1):291-305. doi: 10.1109/TUFFC.2016.2609238. Epub 2016 Sep 13. PMID 27662675
- [Background] White E, Heishman D, Platforms Director S, Che-yi Chao J, Outreach A. Focused Ultrasound Foundation State of the Field 2025 [Internet]. [cited 2025 Nov 19]. Available from: https://cdn.fusfoundation.org/2025/07/31085318/FUSF-State-of-the-Field-2025_July-31.pdf
- [Background] Calik J, Sauer N, Wozniak B, Wojnar A, Pietkiewicz P, Dziegiel P. Pilot Study on High-Intensity Focused Ultrasound (HIFU) for Basal Cell Carcinoma: Effectiveness and Safety. J Clin Med. 2024 Jun 1;13(11):3277. doi: 10.3390/jcm13113277. PMID 38892988
- [Background] Serup J, Bove T, Zawada T, Jessen A, Poli M. High-frequency (20 MHz) high-intensity focused ultrasound: New Treatment of actinic keratosis, basal cell carcinoma, and Kaposi sarcoma. An open-label exploratory study. Skin Res Technol. 2020 Nov;26(6):824-831. doi: 10.1111/srt.12883. Epub 2020 Jun 17. PMID 32557832
- [Background] Al-Jumaily AM, Liaquat H, Paul S. Focused Ultrasound for Dermal Applications. Ultrasound Med Biol. 2024 Jan;50(1):8-17. doi: 10.1016/j.ultrasmedbio.2023.09.004. Epub 2023 Oct 7. PMID 37806924
- [Background] Elhelf IAS, Albahar H, Shah U, Oto A, Cressman E, Almekkawy M. High intensity focused ultrasound: The fundamentals, clinical applications and research trends. Diagn Interv Imaging. 2018 Jun;99(6):349-359. doi: 10.1016/j.diii.2018.03.001. Epub 2018 May 18. PMID 29778401
- [Background] Kuijpers DI, Thissen MR, Berretty PJ, Ideler FH, Nelemans PJ, Neumann MH. Surgical excision versus curettage plus cryosurgery in the treatment of basal cell carcinoma. Dermatol Surg. 2007 May;33(5):579-87. doi: 10.1111/j.1524-4725.2007.33117.x. PMID 17451581
- [Background] Park HE, Park JW, Kim YH, Han JH, Bang CH, Park YM, Lee JH. Analysis on the Effectiveness and Characteristics of Treatment Modalities for Bowen's Disease: An Observational Study. J Clin Med. 2022 May 12;11(10):2741. doi: 10.3390/jcm11102741. PMID 35628868
- [Background] Morton CA, Whitehurst C, Moseley H, McColl JH, Moore JV, Mackie RM. Comparison of photodynamic therapy with cryotherapy in the treatment of Bowen's disease. Br J Dermatol. 1996 Nov;135(5):766-71. PMID 8977678
- [Background] Hernberg Micaela, Mäkelä Siru, Ilmonen Suvi, Vuoristo Mikko, Juteau Susanna, Hannuksela-Svahn Anna, et al. Kansallinen ei-melanoottisten ihosyöpien hoito-ohjeistus. 2025 Dec.
- [Background] WHO, Lucas Robyn, Prüss-Üstün Annette. Solar ultraviolet radiation : global burden of disease from solar ultraviolet radiation. World Health Organization, Public Health and the Environment; 2006.
- [Background] Bentzen J, Kjellberg J, Thorgaard C, Engholm G, Phillip A, Storm HH. Costs of illness for melanoma and nonmelanoma skin cancer in Denmark. Eur J Cancer Prev. 2013 Nov;22(6):569-76. doi: 10.1097/CEJ.0b013e328360150c. PMID 23542376